CLINICAL TRIAL: NCT04126239
Title: Validation Study of a Rapid Screening Test of Food Addiction in Patients Suffering From Obesity and Healthy Volunteer
Brief Title: Validation of a Food Addiction Screening Test
Acronym: FAST - FR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0320
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Food Addiction; Obesity
Keywords: food Addiction; Obesity
MeSH Terms: conditions — Food Addiction; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participant suffering from obesity: Patient, male or female, over 18 and under 70 years old Patient group with a Body Mass Index (BMI) greater than or equal to 30 kg / m2
  Interventions: Other: Online survey - questionnaire
- healthy volunteer
  Interventions: Other: Online survey - questionnaire

INTERVENTIONS:
Other: Online survey - questionnaire — Online survey - questionnaire

SUMMARY:
Food addiction (FA) is a behavioral addiction characterized by a high consumption of palatable foods, which markedly activate the reward system, despite adverse consequences. FA was first described in 1956 but remains controversial. The Yale Food Addiction Scale (YFAS), developed by Gearhardt et al. in 2009, is currently regarded as the "Gold Standard" for FA screening. In a previous study, we established a Food Addiction Screening Test using artificial intelligence. The main objective of the present study is to validate the sensitivity, specificity and precision for FA diagnosis in a sample of patient suffering from obesity and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30
* Able to consent

Exclusion Criteria:

* Non-french speaker
* Patient unable to use internet tools

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * BMI ≥ 30
  * Able to consent
Sampling Method: Non-Probability Sample
Enrollment: 1610 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-10-17 (Estimated); Study Completion 2023-06-17 (Estimated)

PRIMARY OUTCOMES:
FAST score | Baseline
  Screening test to validate
YFAS 2.0 | Baseline
  Screening test to validate DSM-5 Yale Food Addiction Scale (YFAS 2.0)
BES score | Baseline
  Binge Eating Scale scoring
DEBQ score | Baseline
  Dutch Eating Behaviour Questionnaire scoring

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain ICETA, MD, Principal Investigator — Hospices Civils de Lyon; Emmanuel Disse, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France